CLINICAL TRIAL: NCT02352155
Title: Second-look Endoscopy in High Risk Patients After Endoscopic Hemostasis to Their Bleeding Peptic Ulcers Improves Their Outcomes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLOGD
Record Dates: First submitted 2014-12-15; First posted 2015-02-02 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Ulcer Bleeding
Keywords: haemostasis
MeSH Terms: interventions — Epinephrine; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Second look endoscopy (Active Comparator): Second look endoscopy in the following morning with re-treatment to the bleeding vessel using epinephrine injection or heater probe or hemoclips
  Interventions: Procedure: epinephrine injection or heater probe or hemoclips
- observation only (Placebo Comparator): NO second look endoscopy (Observation)
  Interventions: Other: Observation only

INTERVENTIONS:
Procedure: epinephrine injection or heater probe or hemoclips — Elective Second look endoscopy in the following morning with re-treatment to the bleeding vessel using epinephrine injection or heater probe or hemoclips
  Arms: Second look endoscopy
Other: Observation only — Observation for rebleeding, unscheduled endoscopy only when rebleeding criteria fulfilled
  Other Names: Observation for rebleeding
  Arms: observation only

SUMMARY:
Bleeding peptic ulcer is a common medical emergency. Endoscopic treatment stops bleeding in those actively bleeding from their peptic ulcers, reduces further bleeding, transfusion, surgery and deaths. After initial endoscopic control of bleeding, approximately 10% of them will develop recurrent bleeding. Mortality rate in this group of patients is at least 4 fold higher. In the few who need surgery, mortality approaches 30%. Prevention of further bleeding is therefore a major treatment objective. Currently the investigators use a high dose infusion of proton pump inhibitor (PPI) for 72 hours to render gastric pH neutral. In a previous randomized trial, the investigators showed that the rate of bleeding in 30 days was around 7% with such an approach. In a small subgroup of high risk patients defined by presentation with shock and ulcers > 2 cm in size, 1 in 6 would re-bleed. An alternate strategy is to select those at especially high risk of further bleeding and repeat endoscopic treatment the next morning. The investigators have shown that persistence of major bleeding stigmata, i.e. a visible vessel, during a second endoscopy predicts further bleeding. It is therefore logical that by repeating endoscopic treatment the next morning, the investigators can prevent further bleeding and possibly surgery and deaths. The current study proposes to develop a score to identify those at risk of further bleeding after endoscopy. The investigators used a historical cohort with carefully collected clinical data to derive a risk score. In this derivation phase of 939 patients, the investigators have developed a 9 point risk score which consists of the following parameters (Age>60, Male sex, ulcer>2cm, posterior bulbar in location, spurting or Forrest Ia bleeding and admission hemoglobin of < 8 g/dl). Using AUROC and Youden J statistics, a score of 5 or above has been shown to highly predictive of further bleeding. The score will then be validated in a prospective cohort of patients with bleeding peptic ulcers. In the final phase of this study, the investigators propose a randomized controlled trial to test the hypothesis that a second look endoscopy with treatment in selected high risk patients can further reduce bleeding and improve their outcomes. After endoscopic hemostasis to their bleeding peptic ulcers, patients are risk stratified based on the score. Those with a score of 5 or more are randomized to receive the standard treatment (a high dose PPI infusion) or a second look endoscopy with treatment in addition to PPI infusion. The primary outcome to the trial is further significant clinical bleeding.

DETAILED DESCRIPTION:
Hospitalization for bleeding peptic ulcers has declined over past decades [1]. Bleeding from peptic ulcers however remains the commonest diagnosis in those who present with acute upper gastrointestinal bleeding (AUGIB). The incidence has been around 60-80/100,000 population. Endoscopic hemostatic therapy is the first treatment to those with active bleeding and major stigmata of bleeding. Endoscopic therapy stops bleeding and reduces rate of further bleeding, requirement for surgery and importantly deaths [2]. Adjunctive intravenous infusion of a high dose proton pump inhibitor (PPI) further reduces rebleeding. In a multicentre international placebo controlled trial that involved 767 patients with bleeding peptic ulcers, a PPI infusion reduced the rate of further bleeding (10.3 to 5.9% at 72 hour, P=0.026) In a subgroup analysis of a Cochrane meta-analysis over use of PPI in bleeding peptic ulcers, the adjunctive use of PPI in those who underwent endoscopic hemostatic treatment, when compared to those without PPI therapy, was associated with a reduction in deaths (17/954 vs. 32/ 969; OR 0.54; 95%CI 0.3-0.96) [ 4 ] . Despite of aggressive endoscopic therapy and maximal acid suppression using a PPI infusion, further bleeding occurs in around 8% of patients. Further bleeding is the single most important adverse prognostic factor and is associated with a 4 fold increase in mortality. From a National United Kingdom Audit on the management of patients with AUGIB, those who needed surgery for further bleeding and failed endoscopic control had a mortality of 28% [ 5 ]. In addition to initial control of bleeding with endoscopic therapy, the prevention of further bleeding is an important objective.

The use of routine second look endoscopy with re-treatment has been evaluated in several clinical trials. A recent meta-analysis [ 6 ] of these clinical trials concluded that the use of routine second look endoscopy confers a modest reduction in rate of further bleeding. In this pooled analysis of 8 trials and 938 patients, the absolute risk reduction was 6.8% (16.5 to 9.7%). The number to treat to prevent one episode of recurrent bleeding was 15. Only one of these trials used high dose PPI infusion and epinephrine injection alone was used as endoscopic treatment. The use of epinephrine injection is no longer considered an optimal treatment. A second modality should be added to induce vessel thrombosis [ 7 ]. Clinical practice in the reported trials was considered not contemporary. In the modern practice of combination endoscopic treatment and maximal acid suppression, the use of routine second look endoscopy cannot be recommended as the NNT to prevent further bleeding would likely be higher. A policy of routine second look endoscopy is generally not recommended as suggested by an International Consensus Group [ 8 ].

Second look endoscopy in those at high risk of further bleeding is however a logical approach. The NNT to prevent further bleeding diminishes as risk of further bleeding increases. For instance, an ulcer > 2 cm in size with Forrest I or Forrest II a bleeding would be associated with a re-bleeding risk of 15-20% even with high dose PPI infusion. Saeed et al. reported a study consisted of a small number of patients (n=40) and showed that endoscopic re-treatment in selected high risk patients based on a Baylor College score led to significant reduction in further bleeding (0 vs. 24%). This selective approach warrants investigation and could represent a dominant strategy in addition to high dose PPI infusion as a pre-emptive management of patients at high risk of further bleeding. A prerequisite to this approach is a risk score that predicts further bleeding in patients after endoscopic hemostasis and PPI infusion. This risk score needs to be derived from a large cohort of patients after uniform endoscopic treatment and acid suppression. The score will have to be validated in a prospective cohort of patients with bleeding peptic ulcers again after the same aggressive treatment. Furthermore, a randomized controlled trial on the use of second look endoscopy in high risk patients as identified by this risk score is required.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18
* Informed consent obtained
* Successful endoscopic hemostasis
* Risk Score >= 5

Exclusion Criteria:

* Age < 18
* Pregnancy
* Incomplete endoscopic haemostasis -

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2015-02-04 (Actual); Primary Completion 2020-04-02 (Actual); Study Completion 2020-04-02 (Actual)

PRIMARY OUTCOMES:
clinical significant bleeding | 30 days
  1) fresh hematemesis or melena and 2) hypotensive with systolic blood pressure less than or equal to 90 mmHg and pulse rate of greater than or equal to 110 per minute and/ or a drop of haemoglobin of >2g/dl in 24 hours and a hematocrit of 0.24. Further bleeding has to be documented by endoscopic findings or fresh blood in the stomach together with a bleeding or non-bleeding visible vessel.

SECONDARY OUTCOMES:
additional intervention for further bleeding | 30 days
  additional intervention for further bleeding (surgery or angiographic intervention),
blood transfusion | 30 days
  no. of participants with blood transfusion; median blood transfusion
hospitalisation, | 30 days
  hospitalisation (including ICU stay)
treatment related complications | 30 days
  no. of participants with ulcer perforation
deaths from all causes | 30 days
  mortality, (related or not related to treatment ) cause of death

CONTACTS AND LOCATIONS:
Overall Officials: James Y LAU, Prof, Principal Investigator — CUHK
Locations (2):
- Endoscopy Centre, Hong Kong, HONG KONG, China
- Chulalongkorn Memorial Hospital, Bangkok, Pathumwan, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pittayanon R, Suen BY, Kongtub N, Tse YK, Rerknimitr R, Lau JYW. Scheduled second look endoscopy after endoscopic hemostasis to patients with high risk bleeding peptic ulcers: a Randomized Controlled Trial. Surg Endosc. 2022 Sep;36(9):6497-6506. doi: 10.1007/s00464-021-09004-w. Epub 2022 Jan 12. PMID 35020056